CLINICAL TRIAL: NCT01933126
Title: The Effect of HCG Injection to the Uterine Cavity on Pregnancy Rate in Women Undergoing IVF Treatment
Brief Title: Intrauterine Injection of HCG and Implantation Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Assaf Harofeh Medical Center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 151/12
Record Dates: First submitted 2013-02-28; First posted 2013-09-02 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pregnancy Rate; Implantation Rate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCG administration (Experimental): Intrauterine HCG injection
  Interventions: Drug: HCG injection
- Placebo (Placebo Comparator): G2 Medium
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HCG injection
  Arms: HCG administration
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study aims to examine the effect of intrauterine injection of HCG on pregnany rate in women undergoing IVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF treatment

Exclusion Criteria:

* > 40 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Be’er Ya‘aqov, Zerifin, Israel